CLINICAL TRIAL: NCT01239238
Title: Reduction of Asthma Exacerbation Rate in Children by Non-invasive Monitoring of Inflammatory Markers in Exhaled Breath (Condensate): the RASTER Study
Acronym: RASTER
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 10-2-064
Record Dates: First submitted 2010-10-20; First posted 2010-11-11 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Asthma; Children; Home Monitoring; Exhaled Breath Condensate; Non-invasive Inflammatory Markers; Volatile Organic Compounds
Keywords: asthma; children; home monitoring; exhaled breath condensate; non-invasive inflammatory markers; volatile organic compounds
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Care as usual: Therapy is guided based on symptoms and lung function. Assessments: home monitoring, symptoms, lung function, FeNO, asthma control, quality of life and diagnostic assessments of non-invasive inflammatory markers in exhaled air and exhaled breath condensate.

SUMMARY:
The purpose of the present proposal was to investigate the predictive properties of markers in exhaled breath to predict an asthma exacerbation. In addition, the reliability of home monitor assessments to measure asthma control will be examined.

ELIGIBILITY:
Inclusion Criteria:

1. already known with a diagnosis of asthma during at least 6 months
2. age between 6 and 17 years
3. reversibility to a bronchodilator (increase in FEV1 > 9% of predicted value and/or
4. bronchial hyperresponsiveness to histamine < 8 mg/ml.

Exclusion Criteria:

1. cardiac abnormalities
2. mental retardation, congenital abnormalities or existence of a syndrome
3. active smoking
4. no technical satisfactory performance of measurements
5. no phone line or internet assess available at home.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study is carried out in two hospitals in the Netherlands (Maastricht University Medical Centre, Maastricht; and Orbis Medical Centre, Sittard).
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
number of exacerbations | 1 year
  increase of asthma symptoms, use of short b2-agonists, drop in FEV1% of maximum personal value.
asthma control | 1 year
  asthma control questionnaire
Quality of life | 1 year
  Asthma Quality of Life questionnaire for children

SECONDARY OUTCOMES:
cost-effectiveness | 1 year
  incremental cost per exacerbation prevented

CONTACTS AND LOCATIONS:
Overall Officials: Edward Dompeling, PhD MD, Principal Investigator — Maastricht UMC
Locations (2):
- Netherlands (2):
  - Maastricht University Hospital, Maastricht
  - Orbis Medical Centre, Sittard

REFERENCES:
- [Derived] van Vliet D, van Horck M, van de Kant K, Vaassen S, Gulikers S, Winkens B, Rosias P, Heynens J, Muris J, Essers B, Jobsis Q, Dompeling E. Electronic monitoring of symptoms and lung function to assess asthma control in children. Ann Allergy Asthma Immunol. 2014 Sep;113(3):257-262.e1. doi: 10.1016/j.anai.2014.05.015. Epub 2014 Jun 18. PMID 24950912